CLINICAL TRIAL: NCT05825547
Title: Evaluation of Changes in the Immunological Microenvironment Surrounding Subcutaneous Breast Cancer Metastases After Liquid Nitrogen Cryotherapy: Descriptive Pilot Study.
Brief Title: Evaluation of Changes in the Immunological Microenvironment Surrounding Subcutaneous Breast Cancer Metastases After Liquid Nitrogen Cryotherapy
Acronym: CRIMCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EMERGENCE GSO/2020/JF-001
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: cryotherapy; cytotoxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryotherapy (Experimental)
  Interventions: Procedure: Cryotherapy treatment

INTERVENTIONS:
Procedure: Cryotherapy treatment — Cryotherapy treatment administered by an interventional radiologist: the cryotherapy needle is placed under local anesthesia, ultrasound monitoring in real time. A complete cryotherapy cycle is performed with: freezing until the entire tumor is frozen as judged by ultrasound, then thawing for the same duration and refreezing according to the same principle.

SUMMARY:
Cryotherapy is a cold ablation technique used in many tumor locations. The destruction of tissues by cryoablation preserves proteins and in particular anti-tumor antigens, which could induce the stimulation of an immune response. Compared to other interventional radiology techniques, cryotherapy induces a higher immunogenic response. Studies describe complex responses with elevated levels of activating NK cells, circulating and anti-tumor T cells, and pro-inflammatory and NF-KB dependent cytokines.

In breast cancer, whether or not an immune response is triggered depends on the type of cryoablation used. Indeed, high intensity cryoablation (rapid freezing in one cycle of the entire tumor volume) seems to induce a tumor-specific immunodestructive response, whereas low frequency cryoablation (several small repetitive cycles until a sufficient volume of ice is obtained) does not induce an immunogenic response and can even induce an immunoregulation with immunotolerance of the tumor cells The University Hospital of Nîmes has recently acquired a new liquid nitrogen cryotherapy technique, more powerful than the one classically performed with Argon. This technique is used for palliative and analgesic purposes in patients with metastatic breast cancer presenting painful subcutaneous metastases. The aim of this study is to evaluate in these patients the changes in the tumor microenvironment and the immune response potentially induced by this very high intensity cryotherapy.

The study investigators hypothesize that locoregional treatment with liquid nitrogen cryotherapy of subcutaneous breast cancer metastases will allow a systemic response through the induction of an immune response. A better understanding of the type of immune response induced will allow the development of combined therapeutic strategies with curative and not only palliative and analgesic aims.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent
* The patient must be a member or beneficiary of a health insurance plan
* Patient with metastatic breast cancer with painful subcutaneous metastases.
* Patient eligible for cryotherapy.
* Therapeutic decision of antalgic and palliative treatment by cryotherapy taken in Pluridisciplinary Consultation Meeting.
* Patient available for 15-day follow-up.

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study
* The subject us unable to express their consent or refuses to sign the consent form
* The patient is under safeguard of justice or state guardianship

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Description of the immunological makeup of the tumor before liquid nitrogen cryotherapy treatment | Day 0
  Cytometry by Time Of Flight (CyTOF®) mass cytometry analysis of biopsy samples to identify lymphocyte and macrophage populations and anti-tumor markers
Description of the immunological makeup of the tumor after liquid nitrogen cryotherapy treatment | Day 15
  Cytometry by Time Of Flight (CyTOF®) mass cytometry analysis of biopsy samples to identify lymphocyte and macrophage populations and anti-tumor markers

SECONDARY OUTCOMES:
Patients' tolerance to cryotherapy treatment | Day 15
  Collection of complications and adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) criteria
Level of pain related to subcutaneous metastases before cryotherapy treatment | Day 0 immediately before cryotherapy treatment
  0-10 Visual analog scale. Higher scores mean worse outcome.
Level of pain related to subcutaneous metastases after cryotherapy treatment | Day 0 immediately after cryotherapy treatment
  0-10 Visual analog scale. Higher scores mean worse outcome.
Level of pain related to subcutaneous metastases after cryotherapy treatment | Day 15
  0-10 Visual analog scale. Higher scores mean worse outcome.
Pain related to subcutaneous metastases before cryotherapy treatment | Day 0 immediately before cryotherapy treatment
  Brief Pain Inventory (BPI): score from 0-120. Higher scores mean worse outcome.
Pain related to subcutaneous metastases after cryotherapy treatment | Day 0 immediately after cryotherapy treatment
  Brief Pain Inventory (BPI): score from 0-120. Higher scores mean worse outcome.
Pain related to subcutaneous metastases after cryotherapy treatment | Day 15
  Brief Pain Inventory (BPI): score from 0-120. Higher scores mean worse outcome.
Patient reported quality of before cryotherapy treatment | Day 0
  European Organisation for Research and Treatment of Cancer - C30 (EORTC QLQ-C30). This questionnaire is composed of 30 items grouped into 15 scales. A good quality of life is associated with a high score for the functional scales and a low score for the symptom scales
Patient reported quality of after cryotherapy treatment | Day 15
  European Organisation for Research and Treatment of Cancer - C30 (EORTC QLQ-C30). This questionnaire is composed of 30 items grouped into 15 scales. A good quality of life is associated with a high score for the functional scales and a low score for the symptom scales

CONTACTS AND LOCATIONS:
Overall Officials: Julien Frandon, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nimes, Nîmes, France